CLINICAL TRIAL: NCT03849222
Title: Enhancement of Apexification Procedure Outcome of Non Vital Incompletely Formed Roots Using Apical Matrix
Brief Title: Evaluation the Effect of Using of Apical Matrix With Apexification Procedure on Apical Healing of Necrotic Immature Teeth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Maha A Elhussiny , Phd, lecturer of Endodontic in faculty of dentistry Al-Azhar university for girls, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC 61
Record Dates: First submitted 2019-01-04; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Pulp Necrosis; Apexification
Keywords: Open apex; Immature teeth; Non vital pulp; Apical plug; Internal matrix
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Apexification; Pemetrexed; ProRoot MTA

STUDY DESIGN:
Intervention Model Description: participants are allocated at random to receive one of 4 interventions according to the research plan.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ca(OH)2 Apexification (Active Comparator): Apexification was performed with calcium hydroxide. calcium hydroxide dressing was applied directly against the open apex .The canals were back filled with Ca(OH)2 dressing, followed by proper coronal seal. Patients were recalled every 3, 6 and 12 months for evaluation clinically and radiographically. Once the calcific apical barrier was detected the root canals were then obturated and final restoration was done.
  Interventions: Procedure: Apexification; Drug: Ca(OH)2
- Ca(OH)2 Apexification with apical matrix (Experimental): Treated by condensation of calcium hydroxide dressing against an internal matrix , a piece (4X4mm) of resorbable collagen membrane (Biocollagen; Bioteck:Turin, Italy) was gently compacted toward the apex before insertion of Ca(OH)2 dressing, followed by proper coronal seal. Patients were recalled every 3, 6 and 12 months for evaluation clinically and radiographically. Once the calcific apical barrier was detected the root canals were then obturated and final restoration was done.
  Interventions: Procedure: Apexification; Drug: Ca(OH)2; Drug: Apical matrix
- MTA Apexification (Active Comparator): Apexification was performed with MTA as apical plug. A 3-5 mm thickness of MTA using a hand plugger was applied as apical plug and verified radiographically. Moist cotton pellet was placed over the MTA followed by application of coronal seal. After 48 h, the set of the MTA was checked and final obturation of the root canal was done
  Interventions: Procedure: Apexification; Drug: MTA
- MTA Apexification with apical matrix (Experimental): An internal (apical) matrix was used as a base for condensation of MTA apical plug, a pieces of (4X4mm) of resorbable collagen membrane (Biocollagen; Bioteck:Turin, Italy)were compacted toward the apex with premeasured suitable size schilder plugger. Moist cotton pellet was placed over the MTA followed by application of coronal seal. After 48 h, the set of the MTA was checked and final obturation of the root canal was done
  Interventions: Procedure: Apexification; Drug: MTA; Drug: Apical matrix

INTERVENTIONS:
Procedure: Apexification
Drug: MTA
  Other Names: Proroot MTA
  Arms: MTA Apexification; MTA Apexification with apical matrix
Drug: Ca(OH)2
  Other Names: Ca(OH)2 dressing
  Arms: Ca(OH)2 Apexification; Ca(OH)2 Apexification with apical matrix
Drug: Apical matrix — collagen membrane (Biocollagen; Bioteck:Turin, Italy)
  Other Names: internal matrix
  Arms: Ca(OH)2 Apexification with apical matrix; MTA Apexification with apical matrix

SUMMARY:
This study was conducted to evaluate the effect of the use of apical matrix, with Mineral Trioxide Aggregate (MTA) or calcium hydroxide Ca(OH)2 Apexification on apical healing and calcific barrier formation of immature teeth with non- vital pulp.

DETAILED DESCRIPTION:
Conventional root canal ﬁlling procedures are challenging in cases of teeth with necrotic pulp, immature apices, and periapical lesions because of the absence of natural apical constriction and the presence of moisture contamination. In these cases, the risk of extrusion of the root ﬁlling materials and the difﬁculty in managing apical seals compromise the long-term outcome of treatment.

Management of immature teeth with non-vital pulp were confined to custom fitting the filling material, paste fills and apical surgery. The limited success enjoyed by these procedures resulted in significant interest in the phenomenon of establishment of an apical barrier like apexification or continued apical development. Apexification defined as a procedure to induce a calcified barrier in a root with an open apex and necrotic pulp Traditionally, the most commonly used material for apexification is Ca(OH)2 .Despite the high success rate of The long-term Ca(OH)2 apexification , there are several disadvantages to this technique; Length of time for induction of apical hard tissue barriers. Incomplete apical hard tissue barriers because of vascular inclusions.To avoid the challenges associated with long-term Ca(OH)2 apexification procedures, a non-surgical, one-step apexification using MTA as apical plug.

The major problem in cases of a wide open apex is the need to limit the apexification material at the apex, thus avoiding the extrusion of a large amount of material into the periodontal tissue. The use of a matrix is advisable since its placement in the area of bone destruction provides a base on which the sealing material can be packed .

This randomized controlled trial study was carried out to compare the clinical and radiographic outcome of Ca(OH)2 and MTA with or without internal matrix in non-vital immature maxillary incisors.

ELIGIBILITY:
Inclusion Criteria:

* Immature permanent maxillary anterior teeth
* Non vital pulp
* 6-18 years old
* Half or more root length developed Restorable
* No internal or external root resorption
* No horizontal or vertical root fractures
* Fit and healthy patient

Exclusion Criteria:

* Mature
* Vital pulp
* <6 ,>18 years old
* Less than half of the root developed
* Non - restorable
* Root resorption
* Horizontal or vertical root fractures
* Patients with history of uncontrolled diabetes, immunosuppression, severe asthma Patients suffering from periodontal disease

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Change in pain on percussion | baseline, 3 months, 6 months, and 12 months
  Assessed by tapping the tooth with the back of the mirror (Present or absent) binary outcome
Change in swelling and/or sinus | baseline, 3 months, 6 months, and 12 months
  Assessed by visual examination of labial vestibule.The presence of swelling or sinus reported by a binary question yes/no
Change in periapical pathosis | 12 months
  Change in periapical bone density on follow up radiographs to assess the healing process

SECONDARY OUTCOMES:
presence of a calcified apical barrier or not | 3, 6 and 12 months
  Teeth will be reviewed clinically and radiographically in order to detect the calcific barrier formation
Periapical Lesion scored with periapical index ( PAI) | 12 months
  Radio graphically The periapical index provides an ordinal scale of 5 scores ranging from ''healthy'' to ''severe periodontitis with exacerbating features''. (1) Normal periapical structures. (2) Small changes in bone structure. (3) Changes in bone structure with some diffuse mineral loss.(4) Periodontitis with well-deﬁned radiolucent area. (5) Severe periodontitis with exacerbating features. (1, 2: healthy and 3, 4, 5: pathological).baseline, 3 months, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mervat IB Fawzy, Professor, Study Director — Professor of Endodontics AL-Azhar university

IPD SHARING:
Plan to Share IPD: Undecided